CLINICAL TRIAL: NCT04754555
Title: Translation and Transcultural Adaptation of the Arm Activity Measure (ArmA) and Motor Activity Log (MAL) to Assess Perceived Performance of the Upper Limb Use in Adults With Subacute and Chronic Stroke. F-ArmA
Brief Title: Translation and Transcultural Adaptation of the Arm Activity Measure (ArmA) and Motor Activity Log (MAL)
Acronym: F-ArmA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0209
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subacute phase: between 7 days and 6 months post-stroke;
  Interventions: Other: Arm Activity Measure (ArmA) in french
- chronic phase: minimum 6 months post-stroke
  Interventions: Other: Arm Activity Measure (ArmA) in french

INTERVENTIONS:
Other: Arm Activity Measure (ArmA) in french — The Arm Activity Measure (ArmA) provides a standardized assessment of upper limb passive and active perceived performance

SUMMARY:
Upper limb impairment occurs in approximately 70 to 80 per cent of adults post stroke. These impairments will have consequences on functional performance in activities of daily living and hence quality of life. Assessment of upper limb function is a component of rehabilitation that contributes to the selection of optimal interventions according to patient individualized needs. The Arm Activity Measure (ArmA) provides a standardized assessment of upper limb passive and active perceived performance that is only available in it's English version. The aim of this study is to translate and conduct a cross-cultural adaptation of the ArmA is order to investigate its psychometric properties through a validation study among stroke patients.

DETAILED DESCRIPTION:
Assessment of the upper limb post-stroke should be standardized and holistic, representative of multidimensional consequences according the International Classification of Function and Disability (CIF). Measures should demonstrate established psychometric properties, in terms of validity, reproducibility and responsiveness to change. The ArmA allows standardized measurement of both passive and active functions of the upper limb in terms of perceived performance under the activity level of the CIF. To date there is no measure that allows assessment of both upper limb functions of perceived performance in the French language.

Prior to this study, a translation and cross-cultural adaptation (TCCA) of the ArmA was performed in accordance with study objectives and identified gap in the literature. TCCA was conducted in accordance with guidelines for subjective outcome measures contributing to evidence-based practice (Beaton et al., 2000). A six-step translation procedure for self-reported outcome measures was relevant of clinical use in a foreign language. A multidisciplinary team ensured a forwards-backwards translation and cross-cultural adaptation.

An observational, single-center, cross-sectional study design will be implemented to determine the psychometric properties of the French ArmA.

Participants will be from a post-stroke rehabilitation service (as part of their usual care). For the analysis of reliability properties, participants will be hospitalized as part of routine care and participation in the protocol (T0, T1 and T2 assessments) will add 1 to 2 hours of assessment to routine care.

Assessors will be trained Occupational Therapists having participated in the development of the measure.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 with principle diagnosis of first-time ischemic or hemorrhagic stroke at least 7 days since onset and confirmed by MRI or CT;
* participant having returned home from hospitalization at least one night if stroke time since onset is <6 months or resides at home if >6 months since stroke onset;
* participant can maintain attention for questions for at least 30 minutes;
* motivation to participate and having given informed written consent.

Exclusion Criteria:

* subscale of aphasia severity from the Boston Diagnostic Aphasia Examination ≤3 indicating insufficient comprehension and expression for testing;
* subscale score of ≥2 on the agnosia Unilateral Negligence Assessment Battery (BEN) indicating unilateral neglect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with subacute and chronic stroke
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2023-02-09 (Estimated)

PRIMARY OUTCOMES:
Measure OF ArmA inter-rater (test-retest) reproducibility values as measured by intra class coefficients ICC2 | first day of hospitalisation
  The primary outcome measure will be ArmA inter-rater (test-retest) reproducibility values as measured by intra class coefficients ICC2,1.
  Data collection on perceived upper limb performance with the two-step F-ArmA measurement (T0 and T1) will allow the primary outcome (ICC2,1) to be calculated to establish inter-rater reproducibility. ArmA and MAL will be administered on 3 separate occasions by 2 separate assessors.
Measure OF ArmA inter-rater (test-retest) reproducibility values as measured by intra class coefficients ICC2 | 2 to 7 days of first assessment (T0)
  A secondary independent assessor (E2) will assess ArmA and MAL

CONTACTS AND LOCATIONS:
Overall Officials: Claire VILLEPINTE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided